CLINICAL TRIAL: NCT02375100
Title: Comparison of Efficacy of Transversus Abdominis Plane Block and Ilioinguinal Nerve Block for Postoperative Pain Management in Patients Undergoing Inguinal Herniorraphy With Spinal Anesthesia
Brief Title: Transversus Abdominis Plane Block Versus Ilioinguinal Nerve Block for Pain Management in Inguinal Herniorraphy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IzmirBoyaka
Record Dates: First submitted 2015-02-19; First posted 2015-03-02 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Spinal; Acetaminophen; Analgesics; Tramadol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intrathecal bupivacaine&analgesics (Active Comparator): Patients will be given standard care during perioperative period. They will undergo inguinal herniorraphy operation under spinal anesthesia (with 3ml of %0.5 hyperbaric bupivacaine intrathecally) and receive an parenteral pain regimen (acetaminophen for intravenous infusion in two doses routinely and intramuscular tramadol 50 mg when pain score is higher than 4) in postoperative period.
  Interventions: Procedure: Spinal Anesthesia; Drug: Bupivacaine %0.5 (hyperbaric); Device: 25G Quincke needle; Drug: Acetaminophen; Drug: Tramadol
- TAP Block with bupivacaine (Experimental): In addition to standard perioperative care (spinal anesthesia and parenteral pain regimen) patients will receive transversus abdominis plane block (with 20ml of %0.25 isobaric bupivacaine) just before surgery is initiated.
  Interventions: Procedure: Spinal Anesthesia; Procedure: Transversus Abdominis Plane Block; Drug: Bupivacaine %0.5 (hyperbaric); Drug: Bupivacaine %0.25 (isobaric); Device: 25G Quincke needle; Device: Echogenic Needle with 30° bevel; Drug: Acetaminophen; Drug: Tramadol
- IlNB with bupivacaine (Experimental): In addition to standard perioperative care (spinal anesthesia and parenteral pain regimen) patients will receive Ilioinguinal nerve block (with 20ml of %0.25 isobaric bupivacaine) just before surgery is initiated.
  Interventions: Procedure: Spinal Anesthesia; Procedure: Ilioinguinal Nerve Block; Drug: Bupivacaine %0.5 (hyperbaric); Drug: Bupivacaine %0.25 (isobaric); Device: 25G Quincke needle; Device: Echogenic Needle with 30° bevel; Drug: Acetaminophen; Drug: Tramadol

INTERVENTIONS:
Procedure: Spinal Anesthesia — All patients will be administered 3ml of %0.5 bupivacaine through L3-L4 interspace to acquire motor and sensory blockade
  Other Names: Spinal Block
Procedure: Transversus Abdominis Plane Block — Analgesic intervention which will be performed only to Transversus Abdominis Plane Block arm. It requires 20ml of %0.25 bupivacaine administration through a 22 G. x 4 in. (100 mm) Insulated Echogenic Needle with 30° Bevel from midaxillary line between costal margin and anterior superior iliac spine with ultrasound guidance
  Other Names: TAP block
  Arms: TAP Block with bupivacaine
Procedure: Ilioinguinal Nerve Block — Analgesic intervention which will be performed only to Ilioinguinal Nerve Block arm. It requires 10ml of %0.25 bupivacaine administration through a 22 G. x 3-1/8 in. (80 mm) Insulated Echogenic Needle with 30° Bevel between umbilicus and iliac crest where the nerve is detected with ultrasound guidance
  Other Names: IIN Block
  Arms: IlNB with bupivacaine
Drug: Bupivacaine %0.5 (hyperbaric)
  Other Names: Heavy bupivacaine
Drug: Bupivacaine %0.25 (isobaric)
  Other Names: Plain bupivacaine
  Arms: IlNB with bupivacaine; TAP Block with bupivacaine
Device: 25G Quincke needle
Device: Echogenic Needle with 30° bevel
  Arms: IlNB with bupivacaine; TAP Block with bupivacaine
Drug: Acetaminophen — Analgesic drug administration through iv and im route postoperatively. Patients are administered iv acetaminophen 1g twice a day routinely
  Other Names: Analgesics
Drug: Tramadol — Patients will be administered tramadol in postoperative period when their pain score exceeds 4 points (moderate pain)
  Other Names: Analgesics

SUMMARY:
This study compares efficacy of transversus abdominis plane block and ilioinguinal nerve block for postoperative pain in patients undergoing inguinal herniorraphy with spinal anesthesia. One-third of the patients will receive standard postoperative pain regimen(control group), one-third will receive a transversus abdominis plane block (with ultrasound guidance) and the last group will receive an ilioinguinal nerve block(with ultrasound guidance) in addition to standard postoperative pain regimen. This study is a Randomized prospective open-label controlled study.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years old
* having ASA (American Society of Anesthesiologists) 1 or 2 physical status score preoperatively
* not having a neuromuscular disease
* scheduled for elective single sided inguinal herniorraphy operation

Exclusion Criteria:

* being under 18 years of age
* patient refusal
* having a neuromuscular disease or sensorial neurological deficit covering similar area of effect with peripheral nerve block interventions or the surgical site
* having ASA 3 or 4 physical status score preoperatively
* having one of the contraindications to spinal anesthesia and/or to peripheral nerve blocks as listed by NYSORA (New York School of Regional Anesthesia)
* having emergency surgery or scheduled for bilateral inguinal herniorraphy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Pain Assessment with Verbal Descriptor Scale (VDS) | Baseline
Pain Assessment with Verbal Descriptor Scale (VDS) | 2nd hour after surgery
Pain Assessment with Verbal Descriptor Scale (VDS) | 4th hour after surgery
Pain Assessment with Verbal Descriptor Scale (VDS) | 6th hour after surgery
Pain Assessment with Verbal Descriptor Scale (VDS) | 1st day after surgery
Pain Assessment with Verbal Descriptor Scale (VDS) | 2nd day after surgery
Pain Assessment with Verbal Descriptor Scale (VDS) | 1st month after surgery

SECONDARY OUTCOMES:
Complications (Assessment for existence of complications related to procedures in form of Y/N (such as hypotension, bradycardia, arrythmia, hematoma, failed block, nausea, vomiting, urinary retention, headache, back pain)) | Baseline
  Assessment for existence of complications related to procedures (such as hypotension, bradycardia, arrythmia, hematoma, failed block, nausea, vomiting, urinary retention, headache, back pain)
Complications (Assessment for existence of complications related to procedures in form of Y/N (such as hypotension, bradycardia, arrythmia, hematoma, failed block, nausea, vomiting, urinary retention, headache, back pain)) | 2nd hour after surgery
  Assessment for existence of complications related to procedures (such as hypotension, bradycardia, arrythmia, hematoma, failed block, nausea, vomiting, urinary retention, headache, back pain)
Complications (Assessment for existence of complications related to procedures in form of Y/N (such as hypotension, bradycardia, arrythmia, hematoma, failed block, nausea, vomiting, urinary retention, headache, back pain)) | 4th hour after surgery
  Assessment for existence of complications related to procedures (such as hypotension, bradycardia, arrythmia, hematoma, failed block, nausea, vomiting, urinary retention, headache, back pain)
Complications (Assessment for existence of complications related to procedures in form of Y/N (such as hypotension, bradycardia, arrythmia, hematoma, failed block, nausea, vomiting, urinary retention, headache, back pain)) | 6th hour after surgery
  Assessment for existence of complications related to procedures (such as hypotension, bradycardia, arrythmia, hematoma, failed block, nausea, vomiting, urinary retention, headache, back pain)
Complications (Assessment for existence of complications related to procedures in form of Y/N (such as hypotension, bradycardia, arrythmia, hematoma, failed block, nausea, vomiting, urinary retention, headache, back pain)) | 1st day after surgery
  Assessment for existence of complications related to procedures (such as hypotension, bradycardia, arrythmia, hematoma, failed block, nausea, vomiting, urinary retention, headache, back pain)
Complications (Assessment for existence of complications related to procedures in form of Y/N (such as hypotension, bradycardia, arrythmia, hematoma, failed block, nausea, vomiting, urinary retention, headache, back pain)) | 2nd day after surgery
  Assessment for existence of complications related to procedures (such as hypotension, bradycardia, arrythmia, hematoma, failed block, nausea, vomiting, urinary retention, headache, back pain)
Complications (Assessment for existence of complications related to procedures in form of Y/N (such as hypotension, bradycardia, arrythmia, hematoma, failed block, nausea, vomiting, urinary retention, headache, back pain)) | 1st month after surgery
  Assessment for existence of complications related to procedures (such as hypotension, bradycardia, arrythmia, hematoma, failed block, nausea, vomiting, urinary retention, headache, back pain)
First pain perception in postoperative period (The time when the patients experience pain perception after surgery for the first time) | whenever in 48 hours after surgery
  The time when the patients experience pain perception after surgery for the first time
Additional analgesic requirements | Baseline
  Assessment of additional analgesic requirements of patients defined as having a VDS (Verbal Descriptor Scale) greater than 4 (more intense than mild yet lower than moderate)
Additional analgesic requirements | 2nd hour after surgery
  Assessment of additional analgesic requirements of patients defined as having a VDS (Verbal Descriptor Scale) greater than 4 (more intense than mild yet lower than moderate)
Additional analgesic requirements | 4th hour after surgery
  Assessment of additional analgesic requirements of patients defined as having a VDS (Verbal Descriptor Scale) greater than 4 (more intense than mild yet lower than moderate)
Additional analgesic requirements | 6th hour after surgery
  Assessment of additional analgesic requirements of patients defined as having a VDS (Verbal Descriptor Scale) greater than 4 (more intense than mild yet lower than moderate)
Additional analgesic requirements | 1st day after surgery
  Assessment of additional analgesic requirements of patients defined as having a VDS (Verbal Descriptor Scale) greater than 4 (more intense than mild yet lower than moderate)
Additional analgesic requirements | 2nd day after surgery
  Assessment of additional analgesic requirements of patients defined as having a VDS (Verbal Descriptor Scale) greater than 4 (more intense than mild yet lower than moderate)
Additional analgesic requirements | 1st month after surgery
  Assessment of additional analgesic requirements of patients defined as having a VDS (Verbal Descriptor Scale) greater than 4 (more intense than mild yet lower than moderate)

CONTACTS AND LOCATIONS:
Overall Officials: Onur Okur, MD,Resident, Principal Investigator — Izmir Bozyaka Training and Research Hospital
Locations (1):
- Izmir Bozyaka Training and Research Hospital, Izmir, İzmir, Turkey (Türkiye)